CLINICAL TRIAL: NCT00787215
Title: A Survey on the Rate of Glucose Intolerance in Hong Kong Chinese: Validation of the Chinese University Diabetes Screening Score
Brief Title: A Survey on the Rate of Glucose Intolerance in Hong Kong Chinese
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Chair Professor of Medicine and Therapeutics, Chinese University of Hong Kong
Other Study IDs: ADF-2008-3
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes; Impaired Glucose Tolerance (IGT); Impaired Fasting Glucose (IFG); Glucose Intolerance
Keywords: oral glucose tolerance test; Hong Kong Chinese
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- no treatment: observational: no treatment involved
  Interventions: Other: observational: no treatment involved

INTERVENTIONS:
Other: observational: no treatment involved — observational: no treatment involved

SUMMARY:
Hypothesis: There is a high rate of glucose intolerance among Hong Kong Chinese.

The investigators plan to screen Hong Kong Chinese from the community with oral glucose tolerance test (OGTT). The subjects will be referred from GP centers in the community and self-referred with public advertisement on this survey.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese without history of diabetes

Exclusion Criteria:

* known diabetic patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hong Kong Chinese without history of diabetes
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2008-11; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Glucose intolerance status by OGTT | 2 months

SECONDARY OUTCOMES:
Glucose intolerance status predicted by Chinese University Diabetes Risk Score validated by OGTTT | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary Ko, MD, Principal Investigator — Hong Kong Institute of Diabetes and Obesity
Locations (1):
- Gary Ko, Hong Kong, China